CLINICAL TRIAL: NCT03021317
Title: Effects of ACTHAR on Advanced MRI Surrogate Markers of Disease Activity and on Comprehensive Immune Signature During MS Relapses
Acronym: ACTHAR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated early due to lack of resources.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB16-1390
Record Dates: First submitted 2017-01-12; First posted 2017-01-13 (Estimated); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treated Group (Experimental): Open label, single arm treatment study using MRI and laboratory markers to assess efficacy of ACTHAR in MS patients who are undergoing relapses.
  Interventions: Drug: ACTHar

INTERVENTIONS:
Drug: ACTHar — The patients will be given 80 Units subcutaneously of ACTHAR at the time of MS relapse daily for 10 days.
  Other Names: repository corticotropin injection

SUMMARY:
ACTHAR is a FDA approved drug for MS relapses. The purpose of the study is to examine the efficacy of this agent in improving relapses as measured by advanced MRI and laboratory techniques:

1. Advanced serial MRI studies on patients during and after an acute MS relapse. MRI will be performed at baseline, 1 month after the 1st dose of ACTHAR, and months 3, 6, and 12. ACTHAR will be administered for 10 days. Patients will start ACTHAR within 48 hours of relapse assessment.
2. Serial immune assays on patients during and after an acute MS relapse. Serum and blood samples with be collected at baseline, last day of ACTHAR (day 10 of therapy), 1 month post 1st dose, and months 3 and 6.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a demyelinating disease of the CNS. In a vast majority of patients, its clinical course is characterized by transient attacks of acute neurological compromise, followed by variable degree of recovery. Each relapse leaves a patient with some degree of residual disability. Higher number and longer duration of relapses are associated with greater loss of function. Hence, it is imperative that these relapses are optimally treated and curtailed in duration to allow for maximal recovery and repair.

ACTH (ACTHAR or IV formulation) has long been used for the treatment of MS relapses. ACTH has equivalent efficacy to high-dose IV methylprednisolone in curtailing the duration of MS relapses. ACTH has an advantage over steroids in that it has a short half-life and much less deleterious steroid effect on bone and fat metabolism. Importantly, ACTH has a unique mechanism of action on immune and brain cells through melanocortin receptors (MCRs), which promote production of regulatory and anti-inflammatory cytokines and support oligodendrocyte precursors and neuronal function, all of which could lead to better repair of MS lesions and favorable clinical outcome.

The studies proposed herein will provide a better understanding of the effects of ACTHAR in improving MRI lesion characteristics over time. The complementary immune and genetic studies will further provide evidence for the mechanism of action (MOA) of ACTHAR in improving immune dysfunction related to MS relapse. This is a one of a kind study, involving both advanced/state-of-the art MRI techniques and immune studies to assess the beneficial effects of ACTHAR in MS relapses in the same patients over time.

The primary outcome of all MRI techniques is to determine whether there is an improvement and subsequent stabilization/repair over time of tissue damage caused by inflammatory MS disease activity. Multiple conventional and nonconventional MR imaging modalities are examined here to determine which of these are the most sensitive and reliable in detecting microstructural damage and repair over time. The results of this study will also greatly impact the design of future MS trials by providing a guide for selecting the most appropriate MRI and immune methods to assess treatment efficacy in MS.

In terms of laboratory analysis, the following will be examined:

1. Determine immune subset expression in CD4+FOXP3 Tregs and CD8+CD28- T suppressor cells by flow cytometry at each visit.
2. Global gene expression profiling in MNC with 913,000 probes at each visit. Bioinformatics will include pathway analysis and ACTHAR-induced RNA signature.
3. Serum protein profiling for immune-regulated cytokines (Th1, Th2, Th17, monokines…) and neuroprotective proteins (NGF, BDNF, ACTH, HGF, CNTF, IL-10…) at each visit.
4. All data from protein and gene expression, as well as immune subset expression will be compared to our database generated from therapy-naïve stable and exacerbating MS. ACTHAR signature will analyzed based on these comparisons.

ELIGIBILITY:
Inclusion Criteria:

* age > 18
* undergoing a clinical relapse and associated MRI active lesion

Exclusion Criteria:

* Recent infection, any
* use of any glucocorticoid 30 days prior to enrollment
* unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adil Javed, MD, PhD, Principal Investigator — University of Chicago

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants started the trial and received the intervention.
Period: Overall Study
Arm/Group | Treated Group
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: No participants started the trial and received the intervention.
Arm/Group | Treated Group
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous [unit: years]
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment

OUTCOME MEASURES:

1. Primary Outcome: Change in T1 Lesion Relaxation Time
Description: T1 relaxation time is a MRI marker of injury. The change in this metric will be followed over 12 months to see if lesions recover post ACTHAR intervention.
Time Frame: 12 month after the completion of intervention
Population: No participants started the trial and received the intervention.
Arm/Group | Treated Group
Number analyzed (Participants) | 0

2. Secondary Outcome: Change in Immune Subset Expression in CD4+FOXP3 Tregs by Flow Cytometry Post ACTHAR Intervention
Description: Treg cells are unregulated during the healing process in MS relapses. Changes in this population of immune cells will be measured over a course of 6 months post ACTHAR intervention.
Time Frame: 6 month after the completion of intervention
Population: No participants started the trial and received the intervention.
Arm/Group | Treated Group
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed
Arm/Group | Treated Group
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-23): https://cdn.clinicaltrials.gov/large-docs/17/NCT03021317/Prot_SAP_000.pdf
  • Informed Consent Form (2019-10-23): https://cdn.clinicaltrials.gov/large-docs/17/NCT03021317/ICF_001.pdf